CLINICAL TRIAL: NCT01658228
Title: Pilot Combination Treatment Trial of Mild Cognitive Impairment With Depression
Brief Title: Combination Treatment Study for Memory Impairment and Depression
Acronym: DEP-CI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #6459; R01AG040093-01 (NIH)
Record Dates: First submitted 2012-07-30; First posted 2012-08-06 (Estimated); Results first posted 2017-10-17 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Depression; Mild Cognitive Impairment
Keywords: Depression; Dysthymia; Cognitive Impairment; Cognitive Decline; Memory
MeSH Terms: conditions — Depression; Cognitive Dysfunction; Dysthymic Disorder | interventions — Donepezil; Citalopram; Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Donepezil Treatment Group (Other): For the initial 16 weeks of open-label antidepressant treatment, citalopram up to 20 mg daily or venlafaxine up to 225 mg daily was prescribed. At 16 weeks, all patients were randomized, double-blind, to add-on donepezil or placebo for 62 weeks. Donepezil was started at 5 mg and increased to 10 mg daily or maximum tolerated dose while continuing antidepressants.
  Interventions: Drug: Donepezil
- Placebo Treatment Group (Other): For the initial 16 weeks of open-label antidepressant treatment, citalopram up to 20 mg daily or venlafaxine up to 225 mg daily was prescribed. At 16 weeks, all patients were randomized, double-blind, to add-on donepezil or placebo for 62 weeks. Placebo dose was increased during the study to match Donepezil dose increases while continuing antidepressants.
  Interventions: Drug: Placebo
- Citalopram (Other): An open treatment 8 week flexible dosing schedule starting with citalopram 10mg/day for the first week, then increasing to 20 mg/day thereafter to treat the depression. At the week 8 visit, citalopram responders will continue citalopram treatment and will be randomized to add-on donepezil or placebo at the week 16 visit.
  Interventions: Drug: Citalopram
- Venlafaxine (Other): For patients who did not respond to citalopram, open treatment 8 week flexible dosing schedule starting with venlafaxine 37.5mg/day for the first week, then 75mg/day for the second week, then 150mg/day for the third and fourth week, then 225mg/day for the fifth through eighth weeks. At the end of the eighth week, we will assess patients for antidepressant response. At this time-point, venlafaxine responders will be randomized to add-on donepezil or placebo.
  Interventions: Drug: Venlafaxine

INTERVENTIONS:
Drug: Donepezil — Donepezil 5mg will be given for 6 weeks and if tolerated, the dose will be increased to 10 mg per day. The dose range of 5 to 10 mg per day is the recommended dose for donepezil in the treatment of mild to moderate Alzheimer's disease.
  Other Names: Aricept
  Arms: Donepezil Treatment Group
Drug: Placebo — A placebo capsule will be given to randomized subjects for the starting at week 16 and continuing for the remainder of the study. This group will not receive donepezil as treatment.
  Arms: Placebo Treatment Group
Drug: Citalopram — Citalopram tablet will be given to subjects during an 8 week flexible dosing open treatment. If subjects respond to citalopram treatment they will be randomized to add-on donepezil/placebo.
  Arms: Citalopram
Drug: Venlafaxine — Venlafaxine tablet will be given to subjects during an 8 week flexible dosing open treatment if they did not respond to citalopram. If subjects respond to venlafaxine treatment they will be randomized to add-on donepezil/placebo.
  Arms: Venlafaxine

SUMMARY:
Patients presenting with depression (DEP) and cognitive impairment (CI), represent a unique, understudied population that is difficult to diagnose, treat and estimate prognosis. Our pilot data, supported by the literature, suggest that many DEP-CI patients show cognitive decline and often convert to dementia, primarily Alzheimer's disease (AD). In DEP-CI, there is a lack of data on treatment response of mood symptoms to antidepressant treatment and particularly of cognitive deficits to cognitive enhancer treatment. Our initial pilot data in a double-blind study showed that donepezil was superior to placebo in improving memory in antidepressant-treated DEP-CI patients. In a second pilot study, open label es-citalopram plus memantine treatment led to a low rate of conversion to dementia.

In this proposed pilot clinical trial, the investigators will evaluate, treat and follow a broad sample of 80 DEP-CI patients at NYSPI/Columbia University Medical Center (N = 40) and Duke University Medical Center (N = 40). Recruitment will be from clinics and/or advertisements. In the treatment protocol, all 80 DEP-CI patients will receive baseline mood and memory assessments and open antidepressant treatment with citalopram for 8 weeks. At 8 weeks, repeat assessment will occur and patients whose depression has responded to citalopram will be randomized to add-on donepezil or placebo. Non-responders to citalopram will receive open treatment with venlafaxine and will be randomized 8 weeks later (16 weeks of open antidepressant treatment) to add-on donepezil or placebo. Patients will be followed for a total period of 18 months with continuous open antidepressant treatment during the trial.

Donepezil is being studied in order to increase the likelihood of obtaining a signal. If the results are positive, the investigators can begin clarifying the mechanism(s) in subsequent trials. Baseline apolipoprotein E e4 genotype, odor identification deficits, and MRI hippocampal and entorhinal cortex atrophy will be explored as predictors of donepezil response in the 18-month trial. Improving cognition and delaying conversion to a clinical diagnosis of dementia in this high risk group will enhance quality of life, reduce family burden, and markedly diminish overall health care costs.

DETAILED DESCRIPTION:
In the elderly, the most common neuropsychiatric disorders are depression (DEP) and cognitive impairment (CI). Their co-occurrence (DEP-CI) may exceed chance. The lack of research in DEP-CI, the need to determine early prognostic indicators, and to develop optimal treatment strategies, was emphasized by a NIH consensus panel. Since depression in patients with CI increases the risk of conversion to dementia, treatment strategies for DEP-CI have longer-term implications beyond acute antidepressant treatment response. However, in DEP-CI, there is a lack of data on treatment response of mood symptoms to antidepressant treatment and of cognitive deficits to cognitive enhancer treatment, and the long-term prognosis in these patients remains unclear. The investigators have initial pilot data showing that donepezil was superior to placebo in improving memory performance in DEP-CI patients, and pilot data showing that patients with DEP-CI treated with combined escitalopram and memantine have a low conversion rate to dementia, primarily Alzheimer's disease (AD), over one year. This proposal is for the first study to explicitly examine cognitive change, including conversion to dementia, in a randomized, double-blind, placebo-controlled donepezil treatment trial in DEP-CI patients treated openly with antidepressants. The investigators will conduct systematic follow-up to evaluate 18-month outcome. In addition to apolipoprotein E ε4 genotype, the investigators will explore MRI hippocampal and entorhinal cortex atrophy and odor identification deficits as biomarkers that moderate response.

This pilot trial will enroll about 80 DEP-CI patients who present to the departments of Psychiatry, Neurology and Internal Medicine at NYSPI/Columbia University and Duke University medical centers, ensuring broad representation for clinical relevance. In the treatment protocol, all 80 DEP-CI patients will receive open antidepressant treatment with citalopram for 8 weeks. At 8 weeks, citalopram responders will continue to be treated on citalopram, while non-responders will switch to venlafaxine treatment for an additional 8 weeks. At 16 weeks, all subjects will be randomized to add-on donepezil or placebo (N.B. Patients with a prior history of nonresponse to both citalopram and venlafaxine will be enrolled in the protocol and treated with bupropion and subsequently with doctor's choice of antidepressant). Patients will be followed for a total period of up to 18 months in the trial, with antidepressant treatment adjusted as needed based on clinical response and side effects, i.e., open antidepressant treatment is continuous for all subjects throughout the trial and is not the experimental intervention. The investigators chose to study antidepressant plus donepezil compared to placebo based on our pilot data and to increase the likelihood of obtaining a signal.

Aim 1 (primary aim of the study). To assess change in cognitive status over 18 months in antidepressant-treated DEP-CI patients comparing donepezil to placebo.

Hypothesis 1. Antidepressant-treated DEP-CI patients on donepezil will show a lower rate of conversion to dementia, primarily AD, compared to antidepressant-treated DEP-CI patients on placebo by the end of the 18-month trial.

Hypothesis 2 (secondary). Compared to the placebo group, the donepezil group will show better cognitive outcome by the end of the 18-month trial (SRT total recall: primary measure; modified ADAS-cog: secondary measure).

Hypothesis 3 (secondary). At the end of 24 weeks on add-on donepezil or placebo, the donepezil group will show better cognitive outcome than placebo (SRT total recall: primary measure; modified ADAS-cog: secondary measure).

Aim 2: To evaluate moderators of treatment on cognitive change in the 18-month donepezil-placebo trial, based on the view that patients with incipient AD brain pathology will have superior cognitive outcome on donepezil. These Aim 2 hypotheses are considered exploratory.

Hypothesis 1. Patients with the apolipoprotein E ε4 allele (homozygote or heterozygote), compared to patients without this allele, will have better cognitive outcome on donepezil compared to placebo.

Hypothesis 2. Lower scores on the UPSIT (odor identification test) at baseline will be associated with better cognitive outcome on donepezil compared to placebo.

Hypothesis 3. Smaller MRI hippocampal and entorhinal cortex volumes (atrophy) will be associated with better cognitive outcome on donepezil compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Of either sex, age 55-95 years old with minimum 8 years of education who meet criteria for both depression and cognitive impairment as described below.
* Study Criteria for "depression":

  i. Patients who meet DSM-IV symptom criteria for Major Depression or Dysthymia for a minimum of 6 months (2 year duration DSM-IV TR criterion not required for dysthymic disorder in this study). ii. 24-item HAM-D ≥14.
* Study Criteria for "cognitive impairment":

  i. Subjective memory or other cognitive complaints. ii. Score ≤ 11 on the Logical Memory II (Delayed Paragraph Recall, Paragraph A) test from the Wechsler Memory Scale - Revised OR a score that is ≥ 1.5 standard deviations below the norms on the FC SRT
* Folstein Mini Mental State (MMSE) score ≥ 21 out of 30.
* Clinical Dementia Rating (CDR) of 0.5 on the memory item and global rating of 0.5 indicating questionable dementia
* Willing and capable of giving informed consent
* A family member or close friend who consents to serve as informant during the study; this can be a telephone informant in the case of patients who do not have a live-in informant or close significant other.

Exclusion Criteria:

* Meets Criteria for dementia (DSM-IV) or probable Alzheimer's disease (NINCDS-ADRDA criteria)
* Meets DSM IV TR criteria for:

  1. schizophrenia, schizoaffective disorder, psychotic depression or other psychosis, or bipolar I disorder
  2. alcohol or substance dependence or abuse (current or within past 6 months)
* Active suicidal ideation or suicidal attempt in last 6 months.
* Clinical stroke with residual neurological deficits.
* Use of medications known to have a negative impact on cognition: benzodiazepines in lorazepam equivalents ≥ 2 mg daily, narcotics, or anticholinergics. (N.B. Medications that may be associated with cognitive impairment but are rarely considered the likely etiology, e.g, theophylline, nifedipine, Beta blockers, will not be excluded.)
* An acute, severe or unstable medical condition. For cancer, acutely ill patients (including those with metastases) are excluded, but past history of successfully treated cancer does not result in exclusion.
* Presence of any of the following disorders: a) CNS infection, with CSF evidence of meningitis, encephalitis, or other infectious process; b) Post-traumatic dementia, defined as dementia with a clear temporal relationship to a severe head injury where consciousness was lost; c) Huntington's disease; d) Multiple sclerosis; e) Parkinson's disease; f) Other neurologic disorders with focal signs, e.g., amyotrophic lateral sclerosis; g) Mental retardation.
* Contra-indication to MRI scan: pacemaker, metal implants following surgery, any other contraindication to MRI (e.g., ferromagnetic aneurysm clips, heart valves). For patients with possible claustrophobia, they can do the MRI with adjunct lorazepam 0.5 mg to reduce anxiety. Patients who cannot do the MRI scan will still be eligible for the clinical trial, i.e., MRI is optional.

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2011-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davangere Devanand, MD, Principal Investigator — Columbia University; Gregory Pelton, MD, Study Director — Columbia University; Steven Roose, MD, Study Director — Columbia University; Murali Doraiswamy, MD, Study Director — Duke University
Locations (2):
- United States (2):
  - New York State Psychiatric Institute, New York, New York
  - Duke University, Durham, North Carolina

REFERENCES:
- [Derived] Devanand DP, Pelton GH, D'Antonio K, Ciarleglio A, Scodes J, Andrews H, Lunsford J, Beyer JL, Petrella JR, Sneed J, Ciovacco M, Doraiswamy PM. Donepezil Treatment in Patients With Depression and Cognitive Impairment on Stable Antidepressant Treatment: A Randomized Controlled Trial. Am J Geriatr Psychiatry. 2018 Oct;26(10):1050-1060. doi: 10.1016/j.jagp.2018.05.008. Epub 2018 Jun 28. PMID 30037778
- [Derived] Pelton GH, Andrews H, Roose SP, Marcus SM, D'Antonio K, Husn H, Petrella JR, Zannas AS, Doraiswamy PM, Devanand DP. Donepezil treatment of older adults with cognitive impairment and depression (DOTCODE study): clinical rationale and design. Contemp Clin Trials. 2014 Mar;37(2):200-8. doi: 10.1016/j.cct.2013.11.015. Epub 2013 Dec 5. PMID 24315979

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from clinics and/or advertisements.
Pre-assignment Details: 86 subjects were enrolled in the open treatment phase of the study and then 61 subjects were randomized at 16 weeks to the add-on donepezil/placebo treatment groups.
Period: Overall Study
Arm/Group | Donepezil Treatment Group | Placebo Treatment Group
Started | 30 | 31
Completed | 23 | 23
Not Completed | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Donepezil Treatment Group | Placebo Treatment Group | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 6 | 18
  >=65 years | 18 | 25 | 43
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.1 (7.7) | 72.4 (8.9) | 69.8 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 14 | 16 | 30
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 31 | 61

OUTCOME MEASURES:

1. Primary Outcome: Selective Reminding Test (SRT) Total Recall
Description: The 12-item, 6-trial SRT is a memory measure used to assess verbal list learning and memory. The total number of words learned over six trials (total immediate recall) was obtained.
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: Words
Arm/Group | Donepezil Treatment Group | Placebo Treatment Group
Number analyzed (Participants) | 30 | 31
Words | 45.6 (11.2) | 46.6 (11.3)

2. Primary Outcome: Selective Reminding Test (SRT) Delayed Recall
Description: The 12-item, 6-trial SRT is a memory measure used to assess verbal list learning and memory. The total number of words learned over six trials (total immediate recall) and delayed recall (after a 15-minute delay) was obtained.
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: Words
Arm/Group | Donepezil Treatment Group | Placebo Treatment Group
Number analyzed (Participants) | 30 | 31
Words | 7.4 (3) | 7.4 (2.8)

3. Secondary Outcome: Alzheimer's Disease Assessment Scale - Cognitive (ADAS-Cog)
Description: The modified ADAS-Cog is a cognitive battery that assesses learning, memory, language production, language comprehension, constructional praxis, ideational praxis, and orientation. Subjects' scores represent the total number of errors made throughout the various tasks. The total number of possible errors is between 0-85.
Time Frame: Week 16
Measure: Mean (Standard Deviation); unit: number of errors on a scale from 0-85
Arm/Group | Donepezil Treatment Group | Placebo Treatment Group
Number analyzed (Participants) | 30 | 31
number of errors on a scale from 0-85 | 13.2 (6.6) | 13.9 (7.5)

4. Other Pre Specified Outcome: WMS-III Visual Reproduction Subtest
Time Frame: Screen (Week 0), Week 16, Week 40, Week 64, Week 78
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Trails A and B
Description: Parts A and B are composed of 25 circles. Patients are asked to scan the entire page and identify the next number or letter in a sequence.
Time Frame: Screen (Week 0), Week 16, Week 40, Week 64, Week 78
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Stroop
Time Frame: Screen (Week 0), Week 16, Week 40, Week 64, Week 78
Reporting Status: Not Posted

7. Other Pre Specified Outcome: WAIS-III Digit Symbol Subtest
Time Frame: Screen (Week 0), Week 16, Week 40, Week 64, Week 78
Reporting Status: Not Posted

8. Other Pre Specified Outcome: WAIS-III Block Design Subtest
Time Frame: Screen (Week 0), Week 16, Week 40, Week 64, Week 78
Reporting Status: Not Posted

9. Other Pre Specified Outcome: COWAT
Time Frame: Screen (Week 0), Week 16, Week 40, Week 64, Week 78
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Boston Naming
Time Frame: Screen (Week 0), Week 16, Week 40, Week 64, Week 78
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Apolipoprotein E Genotype
Description: Using a standard protocol, DNA is amplified by the polymerase chase reaction (PCR). The genotypes are determined blind to subject status (patient or control) by the sizes of DNA fragments present.
Time Frame: Week 2
Reporting Status: Not Posted

12. Other Pre Specified Outcome: University of Pennsylvania Smell Identification Test (UPSIT)
Description: The subject will "scratch and sniff" 40 common odorants embedded in microcapsules on a separate page. The subject will choose the answer from a 4-item multiple choice list. Scores will range from 0-40.
Time Frame: Screen (Week 0)
Reporting Status: Not Posted

13. Other Pre Specified Outcome: MRI Scan
Description: Images will be obtained using a GE Signa 3 Tesla whole body scanner. T1-weighted sagittal fspgr and T2 FLAIR are the pulse sequences used in order to obtain the MRI images.
Time Frame: Within 1 month of Screen Visit (Week 0)
Reporting Status: Not Posted

14. Other Pre Specified Outcome: WMS-R Logical Memory
Time Frame: Week 0 Screening
Reporting Status: Not Posted

15. Other Pre Specified Outcome: FC-SRT
Time Frame: Week 0 Screening
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Donepezil Treatment Group | Placebo Treatment Group
Serious Adverse Events (participants affected / at risk) | 8/30 | 7/31
Other Adverse Events (participants affected / at risk) | 23/30 | 17/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Donepezil Treatment Group (N=30) | Placebo Treatment Group (N=31)
Cardiac Stents (Cardiac disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2
Allergic Reaction (Immune system disorders) | 1 | 0
Atrial Flutter (Cardiac disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 1
Leg Pain (General disorders) | 0 | 1
Panic Attack (Psychiatric disorders) | 0 | 1
Fugue State (Psychiatric disorders) | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 1
Kidney Stones (Renal and urinary disorders) | 0 | 1
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1
Colorectal Cancer (General disorders) | 1 | 0
Perirectal Abscess (Renal and urinary disorders) | 1 | 0
Right Upper Rotator Cuff Repair (Musculoskeletal and connective tissue disorders) | 1 | 0
Biceps Tendinopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Accidental Injury to Left Arm (Injury, poisoning and procedural complications) | 1 | 0
Stroke (General disorders) | 0 | 1
Parkinson's Disease (Congenital, familial and genetic disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Donepezil Treatment Group (N=30) | Placebo Treatment Group (N=31)
Diarrhea (Metabolism and nutrition disorders) | 12 | 6
Headache/Dizziness (Metabolism and nutrition disorders) | 7 | 5
Upset Stomach (Metabolism and nutrition disorders) | 2 | 2
Nightmares (Psychiatric disorders) | 4 | 2
High Blood Pressure (Cardiac disorders) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 5
Broken Knee (Injury, poisoning and procedural complications) | 0 | 1
Broken 4th Finger (Injury, poisoning and procedural complications) | 0 | 1
Nasal Congestion (General disorders) | 4 | 0
Upper Respiratory Infection (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 1 | 1
Sinus Infection (Infections and infestations) | 1 | 0
Cough (General disorders) | 2 | 0
Restless Leg (Metabolism and nutrition disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 3 | 0
Dry Mouth (General disorders) | 5 | 2
Ear Infection (Infections and infestations) | 1 | 0
Sore Throat (General disorders) | 1 | 1
Pharyngitis (General disorders) | 1 | 0
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Fatigue/Insomnia (General disorders) | 8 | 5
Vomiting (Metabolism and nutrition disorders) | 2 | 1
Constipation (Metabolism and nutrition disorders) | 1 | 2
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Shingles (General disorders) | 1 | 1
Herniated Disk in Neck (Musculoskeletal and connective tissue disorders) | 1 | 0
Poison Ivy (Infections and infestations) | 1 | 2
Fungus on Toes (Infections and infestations) | 1 | 0
Elevated Temperature (General disorders) | 1 | 0
Akathisia (General disorders) | 1 | 0
Unsteadiness (Nervous system disorders) | 1 | 0
GI Reflux (Metabolism and nutrition disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Sweating (General disorders) | 1 | 1
UTI (Renal and urinary disorders) | 2 | 1
Nausea (Metabolism and nutrition disorders) | 3 | 1
Hot Flashes (General disorders) | 1 | 0
Hip Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Weight Loss (Metabolism and nutrition disorders) | 1 | 0
Flu (General disorders) | 1 | 0
Bloating (Metabolism and nutrition disorders) | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1
Vaginal Infection (Infections and infestations) | 0 | 1
Bruxism (General disorders) | 0 | 1
Knee Inflammation (Musculoskeletal and connective tissue disorders) | 0 | 1
Increased Weight (Metabolism and nutrition disorders) | 0 | 1
Increased Appetite (Metabolism and nutrition disorders) | 0 | 1
Flatulence (General disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Lower extremity neuropathy (Nervous system disorders) | 0 | 1
Right Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes